CLINICAL TRIAL: NCT02148809
Title: Blood Volume Analysis of Total Hip Arthroplasty Patients Under Hypotensive Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB # 13193
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Blood Volume Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Volume Analysis, Fluid (Experimental): Preop I-131 is given and the BVA is performed, 6 hours after surgery the same procedure will be done to compare the TBV at both points
  Interventions: Radiation: 1mL of I-131 Human Serum Albumin is injected prior to the measurements

INTERVENTIONS:
Radiation: 1mL of I-131 Human Serum Albumin is injected prior to the measurements

SUMMARY:
Hypotensive Anesthesia is a type of regional anesthesia performed routinely at our hospital. This type of anesthesia reduces the average arterial pressure. Benefits include reduced bleeding and lower risk of blood clots.

The purpose of this study is to determine the effect of intravenous fluids administered with hypotensive anesthesia on your blood volume. With this parameter we will be able to understand how much of your blood is lost because of bleeding and how much of the drop is related to dilution.

Study hypothesis: Hemodilution associated with intravenous fluid substitution during hypotensive anesthesia results in decreased postoperative hemoglobin (Hb) levels

DETAILED DESCRIPTION:
Recent technology allows the measurement of patients' total blood volume with 98% accuracy within 90 minutes or less. This is key to understanding the effect of hypotensive anesthesia on patients undergoing total hip arthroplasty. The drop in blood pressure enhances the dilutional effect of intravenous fluid given during the procedure. Increases in TBV could result in decreases of postoperative hemoglobin. Understanding the effect of hypotensive anesthesia on postoperative hemoglobin levels and TBV will enhance our understanding of postoperative blood management and transfusion triggers.

ELIGIBILITY:
Inclusion Criteria:

* Non- inflammatory degenerative joint disease of the hip
* Patients scheduled for unilateral primary total hip arthroplasty
* Age between 50 and 75 years
* Hypotensive Spinal-epidural anesthesia with systolic BP < 95 and diastolic BP < 65.
* Adequate intraoperative fluid loading: a minimum of 3 L within 6 hours of surgery

Exclusion Criteria:

* Pregnant women or nursing mothers.
* Women of childbearing potential not using adequate birth control methods
* Known hypersensitivity to I-131 albumin or any other component of the Volumex injection kit
* Blood coagulopathies resulting in a hypocoagulable state (hemophilia, von Willebrand disease, etc.)
* Blood coagulopathies resulting in a hypercoagulable state (factor V leiden, antithrombin III deficiency, protein C deficiency, protein S deficiency)
* Patients on anti-coagulants (coumadin, plavix, pradaxa, heparin)
* Congestive Heart Failure (at least one medication to treat congestive heart failure)
* Coronary artery disease (s/p bypass, stent or AMI)
* Kidney insufficiency (creatinine > 1.5)
* Aortic or mitral valve disease
* Pulmonary hypertension
* Revision Hip Surgery
* Inadequate intravenous fluid substitution within the first 6 hrs (<3 liters)
* Inadequate hypotensive anesthesia (mean arterial pressure above 65 for more than 33% of the surgical time

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Niemi TT, Pitkanen M, Syrjala M, Rosenberg PH. Comparison of hypotensive epidural anaesthesia and spinal anaesthesia on blood loss and coagulation during and after total hip arthroplasty. Acta Anaesthesiol Scand. 2000 Apr;44(4):457-64. doi: 10.1034/j.1399-6576.2000.440418.x. PMID 10757582
- [Background] Hahn RG. Haemoglobin dilution from epidural-induced hypotension with and without fluid loading. Acta Anaesthesiol Scand. 1992 Apr;36(3):241-4. doi: 10.1111/j.1399-6576.1992.tb03457.x. PMID 1574972
- [Background] Holte K, Foss NB, Svensen C, Lund C, Madsen JL, Kehlet H. Epidural anesthesia, hypotension, and changes in intravascular volume. Anesthesiology. 2004 Feb;100(2):281-6. doi: 10.1097/00000542-200402000-00016. PMID 14739801
- [Background] Drobin D, Hahn RG. Time course of increased haemodilution in hypotension induced by extradural anaesthesia. Br J Anaesth. 1996 Aug;77(2):223-6. doi: 10.1093/bja/77.2.223. PMID 8881630
- [Background] Manzone TA, Dam HQ, Soltis D, Sagar VV. Blood volume analysis: a new technique and new clinical interest reinvigorate a classic study. J Nucl Med Technol. 2007 Jun;35(2):55-63; quiz 77, 79. doi: 10.2967/jnmt.106.035972. Epub 2007 May 11. PMID 17496003

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Study: 14 patients (7men, 7 women) between 52 and 74 years were enrolled in the study (Table 1).
  Exclusion criteria were blood coagulopathies, medication with anti-coagulants, coronary artery disease, congestive heart failure, kidney insufficiency (creatinine > 1.5 mg/dl), aortic or mitral valve disease, pulmonary hypertension, and known hypersensitivity to the tracer.
  All of them underwent total hip arthroplasty by one high-volume surgeon using a posterior or anterior approach.
Period: Overall Study
Arm/Group | Pilot Study
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Study
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 63.8 [52 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — pilot study with fixed numbers
  Participants
    Female | 7
    Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Blood Volume
Description: The primary outcome is the change in total blood volume (TBV) during the first 6 hours after primary THA utilizing hypotensive anesthesia. Preoperative TBV will be compared to values 6 hours postoperatively.
Time Frame: preoperatively and 6 hours postoperatively
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Pilot Study
Number analyzed (Participants) | 14
ml | 487 (455)

2. Other Pre Specified Outcome: Change IN Plasma Volume PV
Description: An indicator dilution technique was used to measure the blood volume, plasma volume and red cell blood volume. Approved by the Food and Drug Administration in 1998, the BVA-100 blood volume analyzer (Daxor Corp.) is a semi-automated system for blood volume analysis. Prepared standards and injectates were used. The injectate consists of 31I-labeled HSA (370- 1,295 kBq [10-30 mCi]) in saline.
  Measurement was performed directly before surgery in the holding area and 6 hours after surgery.
  Each time, before injection of the tracer a baseline sample was taken. After injection of the tracer via standard i.v. line, the first sample was drawn from an arterial line after 12 minutes waiting time. Afterwards every 6 minutes a sample was taken. In a whole 5 samples were sent for analysis to Daxor® Corp.. Each sample is counted in duplicate.
Time Frame: preoperative and 6 hours postoperatively
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Pilot Study: 14 patients (7men, 7 women) between 52 and 74 years were enrolled in the study
Arm/Group | Pilot Study
Number analyzed (Participants) | 14
ml | 214 (324)

ADVERSE EVENTS:
Time Frame: patients were monitored during length of their hospital stay and at a 4 weeks after surgery follow-up appointment. The Time Frame was 4 weeks.
Arm/Group | Pilot Study
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes